CLINICAL TRIAL: NCT05469958
Title: Efficacy of Perioperative Hypothermia Prevention Measures in Osteosynthesis. Clinical Trial With Control Group and Validation Into Spanish of the "BEDSIDE SHIVERING ASSESSMENT SCALE".
Brief Title: Hypothermia Prevention Measures in Osteosynthesis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, ESther ESpunes Mestres, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021/115-ENF-ASEPEYO nº21/2021; INF-2021-14 (Other: UICatalunya)
Record Dates: First submitted 2022-07-14; First posted 2022-07-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hypothermia; Hypothermia, Accidental; Hypothermia; Anesthesia
Keywords: hypothermia; body temperature; inadvertent hypothermia; unplanned hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Masking Description: It is impossible to mask patients; they will notice whether are warmed or not. The care providers must know which protocol to carry on, so it's impossible to mask them. The PI will prepare the assignation groups by an randomization software.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): a bundle of hypothermia prevention measures will be applied
  Interventions: Other: Hypothermia prevention bundle
- Control group (Active Comparator): Conventional care with textile blankets under patient demand.
  Interventions: Other: Conventional care

INTERVENTIONS:
Other: Hypothermia prevention bundle — pre-warming of the patient for 10 minutes with forced air blankets before the surgery starts, which will be maintained during surgery and during the immediate postoperative period, the intravenous perfusions will be warmed up to 38 Celsius degree (ºC) and the environmental temperature will be controlled at 21 Celsius degree (ºC) during surgery
  Arms: Intervention group
Other: Conventional care — the patient will be attended with textile blankets on patient demand
  Arms: Control group

SUMMARY:
Randomized control study with a control group and 90 days follow-up for assessing the decrease in the incidence of inadvertent perioperative hypothermia in the osteosynthesis surgical patients after the application of a bundle in prevention measures during the perioperative period, assessing thermal comfort, tremors (validation into spanish a tremors assessment scale), surgical site infections and readmissions.

DETAILED DESCRIPTION:
Introduction: Perioperative hypothermia, defined as a core body temperature lower than 36 ºC (Celsius degree), is a major problem in the surgical setting. Between 20 and 70% of patients may develop it unintentionally, affecting, to varying degrees, patient safety. Since the beginning of the 90's, serious complications associated with its appearance have been described: infection, alteration of thermal comfort, shivering and increased readmissions.

Objective: to identify whether the application of a bundle of prevention measures against the occurrence of Inadvertent Perioperative Hypothermia in the osteosynthesis surgical patient decreases the incidence of perioperative hypothermia. Secondary objectives to identify the prevalence of inadvertent perioperative hypothermia in the osteosynthesis surgical patient, to determine if the application of a bundle of preventive measures against the occurrence of inadvertent hypothermia decreases the incidence of postoperative or postanesthetic tremors in the surgical patient, to determine if the application of a bundle of preventive measures against the occurrence of inadvertent hypothermia increases the thermal comfort of surgical patients in the immediate postoperative period, to identify the impact of the application of a bundle of prevention measures against the occurrence of inadvertent perioperative hypothermia in the osteosynthesis surgical patients in relation to surgical site infection up to 90 days postoperative follow up and hospital readmissions associated with the occurrence of infection up to 90 days from surgery, to identify possible variables related to the incidence of surgical site infection at 90 days in the hypothermic patient with respect to the normothermic patient and to validate the Spanish translation of the "BEDSIDE SHIVERING ASSESSMENT SCALE" for tremors in the post anesthesia care unit (PACU).

Methodology:First phase: validation and adaptation to Spanish of the "BEDSIDE SHIVERING ASSESSMENT SCALE" (measurement of tremor in patients) with a prospective study with 40 patients.

Second phase: a controlled Randomized Clinical Trial (RCT) will be carried out, in which the intervention group (IG) will implement the bundle of prevention measures against the appearance of perioperative hypothermia and the control group (CG), the usual treatment with textile blankets will be carried out at the patient's request.

A stratified randomization will be carried out to guarantee an equal distribution by groups in the variables type of operating room, type of anesthesia, anesthetic risk (ASA Physical Status 3, maintaining an equal or similar cluster in both the IG and the CG.

124 osteosynthesis trauma surgery patients will be randomized, 62 in each group.

To the intervention group, a bundle of hypothermia prevention measures will be applied before the start of anesthesia, based on: pre-warming of the patient for 10 minutes with a convective heating system (forced air blankets) which will be maintained during surgery and immediate postoperative period, intravenous perfusions will be warmed to 38 Celsius degree(ºC) and the environmental temperature will be controlled at 21 Celsius degree(ºC) . To the control group, will perform the usual treatment with textile blankets on patient demand as usual.

This study will be carried out at the Economic Health Assistance for Employees and Laborers hospital (ASEPEYO) in Barcelona (Spain) which is an accidents at work hospital. The target population is all patients undergoing osteosynthesis trauma surgery of the upper limb, lower limb, and spine.

Expected results: an improvement in patient safety is expected with a decrease in the incidence of perioperative hypothermia, shivering, with an improvement in postoperative thermal comfort.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing general, spinal locoregional and peripheral locoregional anesthesia, with or without sedation, with nature of elective and urgent surgery in the specialty of trauma surgery with osteosynthesis technique in lower extremities, upper extremities (including clavicle) and spine.

Exclusion Criteria:

* patient in surgical protocol for positive Coronavirus 19 desease, febrile process, thyroid pathology (hypothyroidism/hyperthyroidism), treatment with nitrates, hemodynamically unstable that may require resuscitation with massive intravenous fluids; osteosynthesis in fingers, metacarpals, metatarsals and distal radius fractures, Grade III open fractures, as well as all patients with Quetelet Body Mass Index with value higher than 40 Kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
incidence of perioperative hypothermia | perioperative period (since OR arrival until PACU Discharge)
  Core temperature assessed with 3M (registered trademark) Spot-on dual sensor thermometer. It will be attached to the frontal region of the patient in awake and anesthetized patient. Validated in the USA by Eshragui et al. in 2014. Compared with pulmonary artery catheter (gold standard), difference of 0,5 ºC; validated in Spain by Gómez-Romero et al. in 2019; 289 repeated measures, Spearman correlation coefficient (r) 0.82[95% Confidence Interval (CI)] 0.77-0.85 with p<0.001, with an interrelation coefficient (ICC) of 0.88 (95%CI 0.85-0.90).
  Bland-Altman repeated measures analysis for Spot-On and Swan Ganz catheter revealed a bias (SD) [95% CI] of 0,21°C (0.34) [-2.27 to 2.71].
  Kollmann-Camaiora et al. validated it in 2019 respect to esophageal temperature probe measurement.
  Bland Altman Plot, Pearson Correlation (PC) and intraclass correlation coefficient with 400 repeated measures: PC 0.82, Bias of -0.27(95%CI [-0.61-0.55], and ICC 0.90 (95%CI [0.88-0.92.])

SECONDARY OUTCOMES:
prevalence of inadvertent perioperative hypothermia DESCRIPTION: | perioperative period (since OR arrival until Post Anaesthesia Unit Discharge)
  Core temperature assessed with 3M (registered trademark) Spot-on dual sensor thermometer. It will be attached to the frontal region of the patient in awake and anesthetized patient. Validated in the USA by Eshragui et al. in 2014. Compared with pulmonary artery catheter (gold standard), difference of 0,5 ºC; validated in Spain by Gómez-Romero et al. in 2019; 289 repeated measures, Spearman correlation coefficient (r) 0.82[95% Confidence Interval (CI)] 0.77-0.85 with p<0.001, with an interrelation coefficient (ICC) of 0.88 (95%CI 0.85-0.90).
  Bland-Altman repeated measures analysis for Spot-On and Swan Ganz catheter revealed a bias (SD) [95% CI] of 0,21°C (0.34) [-2.27 to 2.71].
  Kollmann-Camaiora et al. validated it in 2019 respect to esophageal temperature probe measurement.
  Bland Altman Plot, Pearson Correlation (PC) and intraclass correlation coefficient with 400 repeated measures: PC 0.82, Bias of -0.27(95%CI [-0.61-0.55], and ICC 0.90 (95%CI [0.88-0.92.])
incidence of postoperative or postanesthetic tremors in the surgical patient. | postoperative period (since Postanaesthesia care unit arrival until the first documented vital sign registration)
  BEDSIDE SHIVERING ASSESMENT SCALE (BSAS): ordinal scale that evaluates the presence or absence of postoperative or postanesthetic tremors. Created in 2008 by Badjatia et al. it consists of 4 levels, with a minimum value of 0 and a maximum value of 3;
incidence of postoperative or postanesthetic tremors in the surgical patient. assessment of thermal comfort in postanesthesia care unit | postoperative period (since Postanaesthesia care unit (PACU) arrival until PACU discharge)
  Heating, Refrigerating and Air-Conditioning Engineers (ASHRAE) Scale endorsed by the International Organization for Standardization 10551:2019. Scale for measuring indoor thermal comfort.
  It consists of 7 Likert-type items, where the patient is asked the sensation of cold or heat before discharge from the PACU; the center of the scale is thermal neutrality (0), the left pole registers cold, and the minimum score is -3 and the right pole evaluates heat and the maximum value is +3.

OTHER OUTCOMES:
incidence of infection up to 90 days postoperatively. | Data will be collected for the PI three times in the postoperative period; the day 30 after surgery, the day 60 after surgery, and de day 90 after surgery. The day of the surgery will be considered the day 1.
  Self-developed questionnaire created ad-hoc for postoperative data collection (Q2), telephone management: it will be validated in parallel to the clinical research study.
  In relation to infection, the questions will be:
  1. Have you had any wound-related problems such as fluid leakage, positive culture specimen, or spontaneous wound opening after surgery?
  2. Have you required medical follow-up for deliberate opening of the surgical wound?
  3. Have you had localized wound pain, swelling, edema or redness, localized heat, fever?
  4. Have you visited an emergency department because of malaise, feeling of fever or fever higher than 38 Celsius degree(ºC)?
  5. Have you had any imaging test to diagnose infection? The patient will be considered to have infection when an affirmative answer to 3 of the 5 questions is obtained.
incidence of readmission related to infection | Data will be collected for the PI three times in the postoperative period; the day 30 after surgery, the day 60 after surgery, and de day 90 after surgery. The day of the surgery will be considered the day 1.
  Self-developed questionnaire created ad-hoc for postoperative data collection (Q2), telephone management: it will be validated in parallel to the clinical research study.
  In relation to Readmission, the questions will be:
  Have you been readmitted to a hospital for wound-related problems? 7) Have you had surgery to clean the wound in the operating room?

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Gallart Fernández-Puebla, PhD, Study Director — Universitat Internacional de Catalunya; Jordi Castillo Gracía, PhD, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Asepeyo Hospital, Sant Cugat del Vallès, Barcelona-CATALUNYA, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balki I, Khan JS, Staibano P, Duceppe E, Bessissow A, Sloan EN, Morley EE, Thompson AN, Devereaux B, Rojas C, Rojas C, Siddiqui N, Sessler DI, Devereaux PJ. Effect of Perioperative Active Body Surface Warming Systems on Analgesic and Clinical Outcomes: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Anesth Analg. 2020 Nov;131(5):1430-1443. doi: 10.1213/ANE.0000000000005145. PMID 33079867
- [Background] Badjatia N, Strongilis E, Gordon E, Prescutti M, Fernandez L, Fernandez A, Buitrago M, Schmidt JM, Ostapkovich ND, Mayer SA. Metabolic impact of shivering during therapeutic temperature modulation: the Bedside Shivering Assessment Scale. Stroke. 2008 Dec;39(12):3242-7. doi: 10.1161/STROKEAHA.108.523654. Epub 2008 Oct 16. PMID 18927450
- [Background] Kollmann Camaiora A, Brogly N, Alsina E, de Celis I, Huercio I, Gilsanz F. Validation of the Zero-Heat-Flux thermometer (SpotOn(R)) in major gynecological surgery to monitor intraoperative core temperature: a comparative study with esophageal core temperature. Minerva Anestesiol. 2019 Apr;85(4):351-357. doi: 10.23736/S0375-9393.18.12188-2. Epub 2018 Jun 26. PMID 29945430
- [Background] Gomez-Romero FJ, Fernández-Prada M, Fernández-Suárez FE, Gutiérrez-Gonzalez C, Estrada-Martínez M, Cachero-Martínez D, Suárez-Fernández S, García-González N, Picatto-Hernández MD, Martínez- Ortega C, Navarro-Garcia JF. Intra-operative temperatura monitoring with two non-invasive devices (3M SpotOn and Dräger Tcore) in comparison with the swan-Ganz catheter. Cir Cardiov 2019; 26(4): 191-196.
- [Background] Eshraghi Y, Nasr V, Parra-Sanchez I, Van Duren A, Botham M, Santoscoy T, Sessler DI. An evaluation of a zero-heat-flux cutaneous thermometer in cardiac surgical patients. Anesth Analg. 2014 Sep;119(3):543-549. doi: 10.1213/ANE.0000000000000319. PMID 25045862
- [Background] Su SF, Nieh HC. Efficacy of forced-air warming for preventing perioperative hypothermia and related complications in patients undergoing laparoscopic surgery: A randomized controlled trial. Int J Nurs Pract. 2018 Oct;24(5):e12660. doi: 10.1111/ijn.12660. Epub 2018 Apr 23. PMID 29682865
- [Background] Ruetzler K, Kurz A. Consequences of perioperative hypothermia. Handb Clin Neurol. 2018;157:687-697. doi: 10.1016/B978-0-444-64074-1.00041-0. PMID 30459033
- [Background] Granum MN, Kaasby K, Skou ST, Gronkjaer M. Preventing Inadvertent Hypothermia in Patients Undergoing Major Spinal Surgery: A Nonrandomized Controlled Study of Two Different Methods of Preoperative and Intraoperative Warming. J Perianesth Nurs. 2019 Oct;34(5):999-1005. doi: 10.1016/j.jopan.2019.03.004. Epub 2019 Jun 15. PMID 31213348
- [Background] Aydin H, Simsek T, Demiraran Y. Effects of Inadvertent Perioperative Hypothermia on Metabolic and Inflammatory Mediators. Turk J Anaesthesiol Reanim. 2019 Dec;47(6):448-455. doi: 10.5152/TJAR.2019.94715. Epub 2019 Aug 15. PMID 31828241
- [Background] Kang S, Park S. Effect of the ASPAN Guideline on Perioperative Hypothermia Among Patients With Upper Extremity Surgery Under General Anesthesia: A Randomized Controlled Trial. J Perianesth Nurs. 2020 Jun;35(3):298-306. doi: 10.1016/j.jopan.2019.11.004. Epub 2020 Jan 28. PMID 32005604
- [Background] Camus Y, Delva E, Lienhart A. Hypothermie peropératoire non provoquee chez l'adulte. EMC (Elsevier Masson SAS, Paris), Anesthésie-Réanimation, 36-413-A-10,2007.
- [Background] Boddu C, Cushner J, Scuderi GR. Inadvertent Perioperative Hypothermia During Orthopedic Surgery. Am J Orthop (Belle Mead NJ). 2018 Jul;47(7). doi: 10.12788/ajo.2018.0056. PMID 30075036
- [Background] Duff J, Walker K, Edward KL, Ralph N, Giandinoto JA, Alexander K, Gow J, Stephenson J. Effect of a thermal care bundle on the prevention, detection and treatment of perioperative inadvertent hypothermia. J Clin Nurs. 2018 Mar;27(5-6):1239-1249. doi: 10.1111/jocn.14171. Epub 2018 Feb 1. PMID 29149456
- [Background] Nordgren M, Hernborg O, Hamberg A, Sandstrom E, Larsson G, Soderstrom L. The Effectiveness of Four Intervention Methods for Preventing Inadvertent Perioperative Hypothermia During Total Knee or Total Hip Arthroplasty. AORN J. 2020 Mar;111(3):303-312. doi: 10.1002/aorn.12961. PMID 32128778
- [Background] Akers JL, Dupnick AC, Hillman EL, Bauer AG, Kinker LM, Hagedorn Wonder A. Inadvertent Perioperative Hypothermia Risks and Postoperative Complications: A Retrospective Study. AORN J. 2019 Jun;109(6):741-747. doi: 10.1002/aorn.12696. PMID 31135987
- [Background] Scott AV, Stonemetz JL, Wasey JO, Johnson DJ, Rivers RJ, Koch CG, Frank SM. Compliance with Surgical Care Improvement Project for Body Temperature Management (SCIP Inf-10) Is Associated with Improved Clinical Outcomes. Anesthesiology. 2015 Jul;123(1):116-25. doi: 10.1097/ALN.0000000000000681. PMID 25909970
- [Background] Hooper VD, Chard R, Clifford T, Fetzer S, Fossum S, Godden B, Martinez EA, Noble KA, O'Brien D, Odom-Forren J, Peterson C, Ross J, Wilson L; ASPAN. ASPAN's evidence-based clinical practice guideline for the promotion of perioperative normothermia: second edition. J Perianesth Nurs. 2010 Dec;25(6):346-65. doi: 10.1016/j.jopan.2010.10.006. No abstract available. PMID 21126665
- [Background] Duff J, Walker K, Edward K, Williams R, Sutherland-Fraser S. Incidence of Perioperative Inadvertent Hypothermia and compliance with evidence-based recommendations at four Australian hospitals: a retrospective Chart audit. ACORN. 2014; 27(3):16-22.
- [Background] Yi J, Xiang Z, Deng X, Fan T, Fu R, Geng W, Guo R, He N, Li C, Li L, Li M, Li T, Tian M, Wang G, Wang L, Wang T, Wu A, Wu D, Xue X, Xu M, Yang X, Yang Z, Yuan J, Zhao Q, Zhou G, Zuo M, Pan S, Zhan L, Yao M, Huang Y. Incidence of Inadvertent Intraoperative Hypothermia and Its Risk Factors in Patients Undergoing General Anesthesia in Beijing: A Prospective Regional Survey. PLoS One. 2015 Sep 11;10(9):e0136136. doi: 10.1371/journal.pone.0136136. eCollection 2015. PMID 26360773
- [Background] Madrid E, Urrutia G, Roque i Figuls M, Pardo-Hernandez H, Campos JM, Paniagua P, Maestre L, Alonso-Coello P. Active body surface warming systems for preventing complications caused by inadvertent perioperative hypothermia in adults. Cochrane Database Syst Rev. 2016 Apr 21;4(4):CD009016. doi: 10.1002/14651858.CD009016.pub2. PMID 27098439
- [Background] Campbell G, Alderson P, Smith AF, Warttig S. Warming of intravenous and irrigation fluids for preventing inadvertent perioperative hypothermia. Cochrane Database Syst Rev. 2015 Apr 13;2015(4):CD009891. doi: 10.1002/14651858.CD009891.pub2. PMID 25866139
- [Background] Berrios-Torres SI, Umscheid CA, Bratzler DW, Leas B, Stone EC, Kelz RR, Reinke CE, Morgan S, Solomkin JS, Mazuski JE, Dellinger EP, Itani KMF, Berbari EF, Segreti J, Parvizi J, Blanchard J, Allen G, Kluytmans JAJW, Donlan R, Schecter WP; Healthcare Infection Control Practices Advisory Committee. Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017. JAMA Surg. 2017 Aug 1;152(8):784-791. doi: 10.1001/jamasurg.2017.0904. PMID 28467526
- [Background] Carretero-Dios H, Pérez C. Normas para el desarrollo y revisión de estudios instrumentales. Int J Clin Health Psychol.2005; 5(3): 521-551.
- [Background] Carvajal A, Centeno C, Watson R, Martinez M, Rubiales AS. [How is an instrument for measuring health to be validated?]. An Sist Sanit Navar. 2011 Jan-Apr;34(1):63-72. doi: 10.4321/s1137-66272011000100007. Spanish. PMID 21532647
- [Background] Sanchez R, Echeverry J. [Validating scales used for measuring factors in medicine]. Rev Salud Publica (Bogota). 2004 Sep-Dec;6(3):302-18. Spanish. PMID 15656069
- [Background] Matos JR, McSwain JR, Wolf BJ, Doty JW, Wilson SH. Examination of intra-operative core temperature in joint arthroplasty: a single-institution prospective observational study. Int Orthop. 2018 Nov;42(11):2513-2519. doi: 10.1007/s00264-018-3967-y. Epub 2018 May 11. PMID 29752506
- [Background] Rosenberger LH, Politano AD, Sawyer RG. The surgical care improvement project and prevention of post-operative infection, including surgical site infection. Surg Infect (Larchmt). 2011 Jun;12(3):163-8. doi: 10.1089/sur.2010.083. Epub 2011 Jul 18. PMID 21767148
- [Background] Global Guidelines for the Prevention of Surgical Site Infection. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK401132/ PMID 27929621
- [Background] Hypothermia: prevention and management in adults having surgery. London: National Institute for Health and Care Excellence (NICE); 2016 Dec. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK554181/ PMID 32134602
- See also: Spanish Society of Preventive Medicine, Public Health and Hygiene. [Internet].Madrid. Zero Infection Project. — https://infeccionquirurgicazero.es/images/stories/recursos/protocolo/2017/3-1-17-documento-Protocolo-IQZ.pdf
- See also: European Centre for Disease Prevention and Control. [Internet]. Stockholm. Annual reports ECDC. Healthcare-associated infections: surgical site infections. — https://www.ecdc.europa.eu/sites/default/files/documents/AER_for_2017-SSI.pdf
- See also: International organization for standardization (2020). Ergonomics of the thermal environment. (Standard No. 10551:2019. — https://www.iso.org/obp/ui/es/-iso:std:iso:10551:ed-1:v1:en:sec:A

DOCUMENTS (1):
  • Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT05469958/ICF_000.pdf